CLINICAL TRIAL: NCT06559358
Title: Subthreshold Stimulation Versus Suprathreshold Stimulation in People With Chronic Low Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed, Associate Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Beni-Suef University2
Record Dates: First submitted 2024-08-06; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Pain; Trigger Point Pain, Myofascial
MeSH Terms: conditions — Pain; Myofascial Pain Syndromes | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): This group will receive subthreshold stimulation
  Interventions: Device: electrical stimulation
- Group 2 (Experimental): This group will receive suprathreshold stimulation
  Interventions: Device: electrical stimulation
- Group 3 (Sham Comparator): This group will receive no stimulation
  Interventions: Device: electrical stimulation

INTERVENTIONS:
Device: electrical stimulation — A two-channel portable electrical stimulation unit (BTL-4620, Czech Republic).

SUMMARY:
this trial will involve three groups. Group 1 will receive subthreshold stimulation. Group 2 will receive suprathreshold stimulation. Group 3 will receive shame treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 65 years old participated in this study, 2
* Having neck pain for more than 6 months with a grade five or greater on the visual analog scale
* Having one or more trigger points in the upper trapezius muscle,
* A significant increase in neck muscle EMG activity indicates the presence of tender points.

Exclusion Criteria:

* Taking non-pharmacological therapies (e.g., acupuncture, physical therapy, osteopathy)
* Taking oral or intravenous pain therapy, intramuscular or subcutaneous injection of cortisone, or local anesthetics during the study period,
* Presence of any contraindication to electrical current including pregnancy, epilepsy, cardiac arrhythmia, cardiac surgery, implanted pacemaker or defibrillator, previous surgery in the spinal cord, infectious diseases of the spinal cord, malignant tumors with or without secondary blastomas in the spinal cord, severe radicular pain with acute paralysis in the extremities

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2-3 months
  Neck pain intensity will be assessed by the visual analog scale (VAS). Participants will be asked to explain their present pain by putting a mark on a 10 mm horizontal line with 0 degrees indicating "no pain" and 10 indicating the "worst possible pain"
Pressure threshold | 2-3 months
  Myofascial trigger points' sensitivity will be measured by a pressure-pain algometer from upper trapezius muscle.
Electromyography | 2-3 months
  The EMG activity from the upper trapezius muscle will be recorded during rest and voluntary maximum contraction.
Range of motion | 2-3 months
  Flexion, lateral rotation to both sides, lateral flexion to both sides